CLINICAL TRIAL: NCT01570907
Title: A Single Dose, Two-Period, Two-Treatment, Two-Sequence Crossover Bioequivalency Study of Quetiapine Fumarate 25 mg Tablets Under Fasting Conditions
Brief Title: Crossover Bioequivalence Study of Quetiapine Fumarate 25 mg Tablets Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QUET-T25-PVFS-2
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Treatment for Bipolar I Disorder
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Quetiapine Fumarate — 25 mg tablet
  Other Names: Seroquel

SUMMARY:
The objective of this study was to prove the bioequivalence of Roxane Laboratories' Quetiapine Fumarate 25 mg Tablet under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to quetiapine or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States